CLINICAL TRIAL: NCT05868668
Title: Randomized Controlled Trial of Focused Shockwave, Radial Wave, and Sham Therapy for Erectile Dysfunction and Focused Shockwave and Sham Therapy for Chronic Pelvic Pain Syndrome in Patients With and Without History of Prostate Cancer
Brief Title: Efficacy of Low-intensity Shockwave vs Radial Wave for Treatment of Erectile Dysfunction and Pelvic Pain
Acronym: Shockwave
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-103
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction Due to Arterial Insufficiency; Erectile Dysfunction; Erectile Dysfunction Due to Arterial Disease; Chronic Pelvic Pain Syndrome; Chronic Prostatitis; Erectile Dysfunction Following Radical Prostatectomy; Erectile Dysfunction Following Radiation Therapy
Keywords: shockwave; radial wave; pelvic floor physical therapy
MeSH Terms: conditions — Erectile Dysfunction; Spinocerebellar ataxia, autosomal recessive 1

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- fSWT (Experimental): Focused Shock wave treatments
  Interventions: Device: Focused shockwave
- rWT (Active Comparator): Radial wave treatments
  Interventions: Device: Radial wave
- Sham (Sham Comparator): Sham treatments
  Interventions: Device: Sham treatment

INTERVENTIONS:
Device: Focused shockwave — Storz Duolith SD-1 (Storz Medical, Tagerwilen, Switzerland)
  Arms: fSWT
Device: Radial wave — Zimmer enPuls Pro (Zimmer MedizinSysteme GmbH, Neu-Ulm, Germany)
  Arms: rWT
Device: Sham treatment — Handheld sham probe
  Arms: Sham

SUMMARY:
The purpose of this study to perform a randomized, sham controlled analysis of the effectiveness of both fSWT and rWT in the relief of erectile dysfunction and chronic pelvic pain syndrome.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo screening to determine eligibility for study entry. Participants who meet eligibility requirements will be randomized in a double blind manner (participant and investigator) to each treatment arm depending on their primary complaint. Participants with erectile dysfunction will be randomized 2:2:1 to either fSWT, rWT or sham therapy. Patients with chronic pelvic pain syndrome will be randomized 1:1 to either fSWT with pelvic floor physical therapy (PFPT) or PFPT with sham treatment.

ELIGIBILITY:
Erectile Dysfunction Group (ED) Inclusion Criteria (ED): (all of the following)

1. Cis-gendered heterosexual adult males18 years old
2. Stable relationship of more than 3 months duration with currently willing sexual partner and desire for penetration.
3. Mild to moderate organic erectile dysfunction (IIEF-EF score 11-25) in the last 3 months
4. If ED responsive or partially responsive to current use of PDE5I, participant must be willing to discontinue PDE5I for 4 weeks prior to trial and remain off PDE5I for the duration of the study. Partially responsive ED is defined as inadequate response for desired sexual activity, or poorly maintained erection despite initially good response.
5. Agreeable to attempt sexual intercourse at least 4 times per month for duration of study without being under the influence of alcohol or recreational drugs
6. Morning total testosterone level over 300ng/dL

Exclusion Criteria (ED):

1. Nerve-injury related ED (/spinal cord injury, severe lumbosacral disorder (radiculopathy, spinal stenosis) or other neurological disease affecting erectile functions (e.g, multiple sclerosis, alzheimer's disease, parkinsons disease, amyotrophic lateral sclerosis)
2. Untreated hypogonadism (morning total testosterone <300 ng/dL) or on androgen deprivation therapy in the last 12 months
3. Predominately psychogenic ED based upon expert clinician opinion
4. Peyronie's disease, palpable plaque or curvature/penile anatomic abnormality that affects penetrative intercourse to any degree
5. History of non-superficial penile surgery (e.g, penile prosthesis, penectomy, plication, grafting)
6. History of penile injury or trauma (e.g, priapism, penile fracture)
7. Use of intracavernosal injection for ED within the last year
8. If diabetic, HbA1c 8% or higher within the past 12 months
9. Known corporal veno-occlusive dysfunction based on prior Doppler penile ultrasound
10. Current tobacco smoker, or has smoked in the past year
11. Poorly controlled hyperlipidemia
12. Poorly controlled hypertension
13. Severe cardiac disease or history of myocardial infarction
14. History of psychiatric disorder including bipolar disorder, current moderate or severe depression
15. Patients currently using SSRI or psychotropic medication
16. Severe ED based on IIEF-EF (score 10 or below)
17. Current acute prostatitis

Chronic Pelvic Pain Syndrome Group:

Inclusion Criteria (CPPS): (all of the following)

1. Adult males ≥18 years old
2. Chronic pelvic pain not explained by concurrent urinary tract infections. urine)
3. Willing to do PFPT

Exclusion criteria (CPPS):

1. Nerve-injury related pelvic pain (history of /spinal cord injury, severe lumbosacral disorder (radiculopathy, spinal stenosis) or other neurological disease affecting pain in the pelvic region(Multiple sclerosis, Alzheimer's, Parkinsons disease)
2. Acute prostatitis or any acute infection of the pelvic region
3. History of pelvic trauma

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Erectile Dysfunction | baseline, 3 and 6 months
  To evaluate change/minimum clinically important difference (MCID) of International Index of Erectile Function score. Score varies according to baseline ED severity, generally requiring higher value for more severe symptoms.
Chronic Prostatitis/Chronic Pelvic Pain Syndrome: | baseline, 3 and 6 months
  To evaluate change/MCID in Chronic Prostatitis Symptom Index (CPSI) score. Score varies according to baseline ED severity, generally requiring higher value for more severe symptoms.

SECONDARY OUTCOMES:
Erectile Dysfunction | baseline, 3 and 6 months
  SEP- Sexual Encounter Profile Questionnaire (log diary 5-item questionnaire with yes/no questions after sexual attempt)
Erectile Dysfunction | baseline, 3 and 6 months
  GAQ- Global Assessment Questionnaire. Two yes/no questions assessing for improvement in sexual function.
Erectile Dysfunction | baseline, 3 and 6 months
  EHS- Erection Hardness Score measuring erection hardness with a higher score indicating more rigidity.

CONTACTS AND LOCATIONS:
Overall Officials: Petar Bajic, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No